CLINICAL TRIAL: NCT04278729
Title: A Prospective Multi-dose Study of Apixaban in Subjects With Nephrotic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2233
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Nephrotic Syndrome; Membranous Nephropathy
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulonephritis, Membranous | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nephrotic Syndrome Arm (Experimental): Patients diagnosed with Nephrotic syndrome will be in this arm.
  Interventions: Drug: Apixaban 5 MG
- Healthy Arm (Experimental): Healthy volunteers will be in this arm.
  Interventions: Drug: Apixaban 5 MG

INTERVENTIONS:
Drug: Apixaban 5 MG — 1 - 5 mg tablet taken orally twice a day
  Other Names: Eliquis

SUMMARY:
This phase I study is a single arm, multi-dose study that will evaluate steady-state apixaban pharmacokinetics (PK) and pharmacodynamics (PD) in subjects with Nephrotic Syndrome (NS) vs healthy control subjects. This study will enroll 20 subjects diagnosed with NS and 10 healthy control subjects. Comparing differences in steady-state apixaban PK/PD parameters between subjects with NS and healthy volunteers will be essential to identifying a safe and effective apixaban dose and dose administration schedule for future randomized controlled trials (RCTs).

ELIGIBILITY:
Inclusion Criteria:

Study Subjects

* 18-79 years of age
* Confirmed diagnosis of NS, with at least one of the following (confirmed within 1 month prior to scheduled Day 1 Study Visit):
* Nephrotic-range proteinuria, defined as >3.0 g/24 hours
* UPC (ratio of protein to creatinine in random spot urine sample), defined as >3.0
* Hypoalbuminemia, defined as <3.0 g/dL

Control Subjects

* 18-79 years of age
* Normal albumin levels (>3.0 mg/dL)
* No history of chronic kidney disease

Exclusion Criteria:

* Age <18 or ≥80 years old
* Serum Creatinine (SCr) ≥1.5 AND weight ≤60kg (these subjects would receive a reduced apixaban dose, per drug labeling)
* Weight >120 kg OR body mass index (BMI) ≥40 kg/m^2
* Estimated Glomerular Filtration Rate (eGFR) <15 mL/min or on dialysis
* Signs and symptoms of increased risk of bleeding, including but not limited to: frequent nosebleeds, unexplained or worsening bruising, blood in urine or stool
* Unwilling to avoid engaging in activities that may increase the risk of bleeding through body injury or bruising, during the study period (e.g., contact sports)
* Baseline prolonged INR, defined as INR >1.4

  * If INR is elevated, but PT and aPTT are below the upper limit of normal (13.3 sec and 37.7 sec, respectively), then the subject may be cleared to receive the study drug at the discretion of one of the study physicians.
* Platelets <100 x 109/L
* History of stroke, or a history of gastrointestinal or intracranial bleeds
* Use of any prescription medications, over-the-counter (OTC) medications, or herbal products that are strong inhibitors or inducers of CYP3A4 and/or P-gp within 14 days prior to Study Day 1 or anticipated need for such drugs during the study. Examples included:

  * Strong inducers of CYP3A4 (e.g., rifampin, carbamazepine, phenytoin, St. John's Wort, etc.)
  * Strong inhibitors of CYP3A4 (e.g., ketoconazole, ritonavir, clarithromycin, etc.)
  * Antiplatelet and/or anticoagulant agents: heparin, aspirin** (see below), clopidogrel, prasugrel, non-steroidal anti-inflammatory drugs (NSAIDs), warfarin, rivaroxaban, dabigatran, edoxaban
* Pregnancy or breastfeeding
* Liver disease with impaired synthetic function (INR >1.4, total bilirubin >1.2)
* Evidence of acute kidney disease by the KDIGO criteria (>1.5 x baseline SCr, or >0.3 mg/dL increase in SCr, over past 48 hours
* Unwillingness to forgo drinking alcohol during the study period due to heightened bleeding risk.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Steady-state Area Under the Plasma Concentration Versus Time Curve From Time Zero to 12 Hours of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Area Under the Curve (AUC (0-12)) is the area under the curve from time 0 to 12 hour after apixaban steady state concentration is reached.

SECONDARY OUTCOMES:
Initial Dose Area Under the Plasma Concentration Versus Time Curve From Time Zero to 12 Hours of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  AUC (0-12) is the area under the curve from time 0 to 12 hour after the initial dose
Steady state Elimination of Half-Life of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Mean terminal phase plasma t½ of apixaban at steady-state
Initial dose Elimination of Half-Life of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Mean terminal phase plasma t½ of apixaban after initial dose
Steady-state Maximum Observed Plasma Concentration of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Maximum observed drug concentration in plasma after administration (Cmax) of apixaban at steady-state
Initial dose Maximum Observed Plasma Concentration of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Maximum observed drug concentration in plasma after administration (Cmax) of apixaban after initial dose
Steady state Plasma Clearance as a Function of Bioavailability of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  CL/F of apixaban of apixaban at steady-state
Initial dose Plasma Clearance (CL) as a Function of Bioavailability (F) of Apixaban | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  CL/F of apixaban of apixaban after initial dose
Initial Thrombin Generation Assay (TGA) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Initial apixaban TGA concentrations. Thrombin generation assay is used to investigate hypo- or hypercoagulability.
Steady state Thrombin Generation Assay (TGA) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Steady state apixaban TGA concentrations. Thrombin generation assay is used to investigate hypo- or hypercoagulability.
Initial dose Anti-Xa activity | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Initial apixaban dose Anti-Xa activity. Anti-Xa activity will be used to measure plasma apixaban levels.
Steady state Anti-Xa activity | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Steady state apixaban dose Anti-Xa activity. Anti-Xa activity will be used to measure plasma apixaban levels.
Initial dose Activated Partial Thromboplastin Time (aPTT) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Initial apixaban dose aPTT. The activated partial thromboplastin time (aPTT) will be used to characterize the coagulation of the blood.
Steady state Activated Partial Thromboplastin Time (aPTT) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Steady state apixaban dose aPTT. The activated partial thromboplastin time (aPTT) will be used to characterize the coagulation of the blood.
Initial dose International Normalised Ratio (INR) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Initial apixaban dose INR. INR is defined as the ratio of the participants prothrombin time and the normal mean prothrombin time. The INR will help determine the risk of coagulation.
Steady state International Normalised Ratio (INR) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Steady state apixaban dose INR. INR is defined as the ratio of the participants prothrombin time and the normal mean prothrombin time. The INR will help determine the risk of coagulation.
Initial dose Prothrombin time (PT) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose
  Initial apixaban dose PT. Prothrombin is defined as time taken by the blood to clot in the participants.
Steady state Prothrombin time (PT) | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 8
  Steady state apixaban dose PT. Prothrombin is defined as time taken by the blood to clot in the participants.
Total Adverse Events (AE) | From screening to Day 10 after initial study drug administration
  Number of subjects experiencing AEs, bleeding-related AEs, serious adverse events (SAEs), or discontinuations due to AEs

OTHER OUTCOMES:
Pharmacogenetics and AUC0-12 | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 1 & 8
  Associations between germline variants within genes that encode proteins that are central to apixaban metabolism and transport and AUC0-12
Pharmacogenetics and CL/F | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 1 & 8
  Associations between germline variants within genes that encode proteins that are central to apixaban metabolism and transport and CL/F
Pharmacogenetics and t1/2 | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 1 & 8
  Associations between germline variants within genes that encode proteins that are central to apixaban metabolism and transport and t1/2
Pharmacogenetics and anti-Xa | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 1 & 8
  Associations between germline variants within genes that encode proteins that are central to apixaban metabolism and transport and anti-Xa
Pharmacogenetics and thrombin generation | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 1 & 8
  Associations between germline variants within genes that encode proteins that are central to apixaban metabolism and transport and thrombin generation
Pharmacogenetics and Cmax | Predose; 1, 2, 3, 4, 6, and 8 hours (hr) postdose approximately on Day 1 & 8
  Associations between germline variants within genes that encode proteins that are central to apixaban metabolism and transport and Cmax
Baseline Quantitative D-Dimer | Baseline at hour 0
  Quantitative D-Dimer levels at baseline before first dose of apixaban
Quantitative D-Dimer at steady-state | Day 8 at hour 8
  Quantitative D-Dimer levels at steady-state apixaban

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Crona, PharmD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No